CLINICAL TRIAL: NCT05231265
Title: Effect of Lumbar Surgery on Complexity During a Walking Task in the Chronic Low Back Pain Patient
Brief Title: Effect of Lumbar Surgery on Complexity During a Walking Task in Chronic Low Back Pain
Acronym: LOBAFRACS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-2/AH-2
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Low Back Pain
  Interventions: Other: Walking task

INTERVENTIONS:
Other: Walking task — Treadmill walking task with study of fractal variability (complexity) for 10 minutes.

SUMMARY:
Lumbar surgery is the most common treatment for chronic disabling low back pain with degenerative disc disease. There are few elements to objectively evaluate the improvement of the motor control after surgery and the motor adaptation capacities of the patients.

The impact of lumbar surgery on complexity in this painful context has never been studied. Theoretically, the restriction of mobility imposed by lumbar surgery should limit the subject's adaptive capacities (of one or more lumbar segments) and thus reduce complexity. Nevertheless, improvement in pain intensity levels could allow the patient to find better motor adaptation capacities, necessary for a positive evolution in the long-term.

The aim of this study was to investigate the evolution of gait complexity in chronic low back pain patients pre- and post-surgery. If surgery improves the adaptability of walking through an antalgic benefit exceeding the induced stiffness, the complexity of walking should be superior after surgery.

This is a proof-of-concept study in which the study investigators hypothesize that measuring complexity by fractal analysis during a walking task will show the increase in gait complexity induced by lumbar surgery at 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain requiring prosthesis or arthrodesis surgery on one or two levels
* Subject affiliated or beneficiary of a health insurance plan.
* The patient must have given their free and informed consent

Exclusion Criteria:

* Patients with organic low back pain (infection, tumor, inflammatory rheumatism)
* Patient with a neurological deficit (cauda equina syndrome or motor testing MRC < 3 on a muscle group of the lower limbs)
* Patient who has already undergone lumbar surgery (except single discectomy)
* Patient with serious concomitant pathologies
* Patients participating in a therapeutic study prohibiting participation in another study
* Patient in an exclusion period from a different study
* It is impossible to give the subject informed information
* Patient is unable to express consent
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain requiring prosthesis or arthrodesis surgery for their lumbar pathology (surgery on one or two levels) followed at the Nîmes University Hospital or at the Grand Sud Polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Gait complexity | 10 days before surgery +/- 3 days
  fractal analysis of gait variability: value normally between 0.5 (degraded structure) to 1 (optimal structure)
Gait complexity | Month 3
  fractal analysis of gait variability: value normally between 0.5 (degraded structure) to 1 (optimal structure)
Gait complexity | Month 6
  fractal analysis of gait variability: value normally between 0.5 (degraded structure) to 1 (optimal structure)

SECONDARY OUTCOMES:
Patient reported pain | 10 days before surgery +/- 3 days
  Visual analog scale (0-100)
Patient reported pain | Month 3
  Visual analog scale (0-100)
Patient reported pain | Month 6
  Visual analog scale (0-100)
Apprehension of pain of movement | 10 days before surgery +/- 3 days
  Tampa Scale of Kinesiophobia. Score ranging from 17-68. Higher scores denote greater level of kinesiophobia (a score >40 is considered significant kinesiophobia)
Apprehension of pain of movement | Month 3
  Tampa Scale of Kinesiophobia. Score ranging from 17-68. Higher scores denote greater level of kinesiophobia (a score >40 is considered significant kinesiophobia)
Apprehension of pain of movement | Month 6
  Tampa Scale of Kinesiophobia. Score ranging from 17-68. Higher scores denote greater level of kinesiophobia (a score >40 is considered significant kinesiophobia)
Patient reported quality of life | 10 days before surgery +/- 3 days
  EuroQol-5 Dimension questionnaire: results generated as 5 digit number corresponding to different aspects of quality of life
Patient reported quality of life | Month 3
  EuroQol-5 Dimension questionnaire: results generated as 5 digit number corresponding to different aspects of quality of life
Patient reported quality of life | Month 6
  EuroQol-5 Dimension questionnaire: results generated as 5 digit number corresponding to different aspects of quality of life
Correlation between type of surgery and gait variability | 10 days before surgery +/- 3 days
  Classified as either arthrodesis or prosthesis
Correlation between type of surgery and gait variability | Month 3
  Classified as either arthrodesis or prosthesis
Correlation between type of surgery and gait variability | Month 6
  Classified as either arthrodesis or prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Homs, Principal Investigator — CHU Nimes
Locations (2):
- France (2):
  - CHU Nîmes, Nîmes
  - Polyclinique Grand Sud, Nîmes

IPD SHARING:
Plan to Share IPD: No